CLINICAL TRIAL: NCT04783844
Title: Usefulness of 3D Digital Reconstruction in the Imaging Diagnosis of Pancreatic Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, David Ferreras, Principal Investigator, Hospital Universitario Virgen de la Arrixaca
Other Study IDs: Virtual pancreas
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Pancreas Neoplasm
Keywords: 3D virtual model
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Virtual modelization. — 3D-MSP technology is used to make virtual 3D models based on conventional CT.

SUMMARY:
Reconstruction using 3D virtual models has brought about a revolution in diagnostic imaging and its use is increasingly widespread. The objective of this work is to determine the precision of the 3D model when establishing the characteristics of tumors and their relationship with other anatomical structures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected pancreatic tumor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected pancreatic tumor.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 1 day
  To evaluate the correlation between the findings in the virtual model and in the CT.

CONTACTS AND LOCATIONS:
Locations (1):
- David Ferreras, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No